CLINICAL TRIAL: NCT02860676
Title: A Phase 1 Extension Study to Determine the Safety of UC-961 (Cirmtuzumab) at the Recommended Phase 2 Dose for Retreatment of Patients With Chronic Lymphocytic Leukemia Treated Previously With UC-961
Brief Title: Extension Study of UC-961 (Cirmtuzumab) for Patients With Chronic Lymphocytic Leukemia Treated Previously With UC-961
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Catriona Jamieson, Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150851
Record Dates: First submitted 2016-06-09; First posted 2016-08-09 (Estimated); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; cancer; UC-961; cirmtuzumab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms | interventions — cirmtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cirmtuzumab (Experimental): Cirmtuzumab 16 mg/kg administered every 14 days for 4 doses, then every 28 days for 4 doses via intravenous infusion.
  Interventions: Drug: cirmtuzumab

INTERVENTIONS:
Drug: cirmtuzumab
  Other Names: UC-961

SUMMARY:
The purpose of the study is to investigate the safety of the investigational drug called cirmtuzumab when given for a duration of 6 to 12 months. Cirmtuzumab is a type of drug called a monoclonal antibody. This drug is designed to attach to a protein called ROR1 that is on the surface of chronic lymphocytic leukemia (CLL) cells. This blocks growth and survival of the CLL cells. ROR1 is rarely expressed on healthy cells so this drug should target the cancer cells. Cirmtuzumab is considered experimental because its use is not approved by United States (US) Food and Drug Administration (FDA).

Although there is evidence from tests on laboratory animals that cirmtuzumab can decrease the number of CLL cells, the investigators do not know if this will work in humans. Therefore, the goal of this study is to see if cirmtuzumab is safe and tolerable in study participants when given for a duration of 6 to 12 months.

DETAILED DESCRIPTION:
This is an open-label extension study to determine the safety and tolerability of cirmtuzumab given to participants who enrolled and completed the initial phase 1 trial in CLL without a dose-limiting toxicity.

UC-961 is administered by intravenous infusion every 14 days for 4 doses, then every 28 days for 4 doses, after which responses will be assessed. Patients with an objective response (meeting working group criteria for partial response or complete response) will continue at the same dose and schema. Patients with stable disease or progressive disease are eligible to increase the dose of UC-961 for another 6-month course.

Duration of UC-961 administration is until disease progression, treatment intolerance, or lack of clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and phenotypic verification of B cell CLL and measurable disease. Immunophenotyping of the leukemic cells (blood or marrow) must demonstrate a monoclonal (or light chain positive) B cell population with immunophenotype consistent with CLL (e.g., co-expressing CD19 and CD5).
* Recovered from toxic effects attributed to UC-961 to grade 1 levels, or baseline.
* Must have measurable disease, including one of the following:

  * absolute lymphocyte count greater than 5000/microliter
  * lymphadenopathy greater than 1.5 cm in longest dimension
  * splenomegaly
  * bone marrow biopsy with residual CLL cells, or resultant bone marrow dysfunction
* Women of childbearing potential must agree not to become pregnant for the duration of the study. Both men and women must agree to use a barrier method of contraception for the duration of the study and until 10 weeks after the final dose of UC-961.
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Adequate hematologic function
* Adequate renal function
* Adequate hepatic function
* Adequate coagulation tests

Exclusion Criteria:

* Pregnant or breast-feeding women
* May have had intervening therapy since completion of initial UC-961 dosing, but excluding the following:

  * Within 7 days of UC-961 restart, or 5 half-lives (if known), whichever is shorter: small molecule tyrosine kinase inhibitor (eg: ibrutinib, idelalisib, AVL-292, IPI-145);
  * Within 28 days of UC-961 restart: chemotherapy (e.g., purine analogues, alkylating agents), corticosteroids, radiation therapy, or participation in any other investigational drug treatment (besides UC-961);
  * Within 56 days of UC-961 restart: previous UC-961 dosing;
  * Within 56 days of UC-961 restart: monoclonal antibody therapy directed against CLL (e.g., rituximab, ofatumumab, obinutuzumab, alemtuzumab).
* Current infection requiring parenteral antibiotics.
* Active infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
* Concurrent malignancy or prior malignancy within the previous 3 years (other than completely resected carcinoma in situ, prostate cancer, or localized non-melanoma skin cancer).
* Known central nervous system (CNS) involvement by malignancy.
* Untreated autoimmunity such as autoimmune hemolytic anemia, or immune thrombocytopenia.
* Uncompensated hypothyroidism (defined as thyroid stimulating hormone greater than 2x upper limit of normal not treated with replacement hormone).
* Presence of more than 55% pro-lymphocytes in peripheral blood. Patients with Richter's transformation are not excluded.
* Insufficient recovery from surgical-related trauma or wound healing.
* Impaired cardiac function including any of the following:

  * Myocardial infarction within 6 months of starting study drug;
  * A past medical history of clinically significant electrocardiogram (ECG) abnormalities;
  * Other clinically significant heart disease (e.g. uncontrolled congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catriona Jamieson, MD, PhD, Principal Investigator — University of California, San Diego; Michael Y Choi, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States

REFERENCES:
- [Background] Choi MY, Widhopf GF 2nd, Ghia EM, Kidwell RL, Hasan MK, Yu J, Rassenti LZ, Chen L, Chen Y, Pittman E, Pu M, Messer K, Prussak CE, Castro JE, Jamieson C, Kipps TJ. Phase I Trial: Cirmtuzumab Inhibits ROR1 Signaling and Stemness Signatures in Patients with Chronic Lymphocytic Leukemia. Cell Stem Cell. 2018 Jun 1;22(6):951-959.e3. doi: 10.1016/j.stem.2018.05.018. PMID 29859176

RESULTS

PARTICIPANT FLOW:
Groups:
- Cirmtuzumab: Cirmtuzumab 16 mg/kg
Period: Overall Study
Arm/Group | Cirmtuzumab
Started | 3
Completed | 2
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cirmtuzumab
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-emergent Adverse Events as Assessed by CTCAE v4.0
Description: Adverse events (AE) assessed by CTCAE v4.0 during cirmtuzumab treatment and during 3 months of follow-up
Time Frame: From start of investigational treatment to discontinuation from trial participation, on average 159 days
Measure: Number; unit: Adverse Events
Groups:
- Grade 1 Adverse Events: Number of CTCAE Grade 1 adverse events among all study subjects
- Grade 2 Adverse Events: Number of CTCAE Grade 2 adverse events among all study subjects
- Grade 3 Adverse Events: Number of CTCAE Grade 3 adverse events among all study subjects
- Grade 4 Adverse Events: Number of CTCAE Grade 4 adverse events among all study subjects
Arm/Group | Grade 1 Adverse Events | Grade 2 Adverse Events | Grade 3 Adverse Events | Grade 4 Adverse Events
Number analyzed (Participants) | 3 | 3 | 3 | 3
Adverse Events
  Eye disorders | 1 | 0 | 0 | 0
  Abdominal pain | 1 | 0 | 0 | 0
  Constipation | 0 | 1 | 0 | 0
  Gastrointestinal disorders, other | 0 | 1 | 0 | 0
  Dizziness | 2 | 0 | 0 | 0
  Upper respiratory infection | 0 | 1 | 0 | 0
  Generalized muscle weakness | 1 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders, other | 1 | 0 | 0 | 0
  Thrombocytopenia | 7 | 0 | 0 | 0
  Anemia | 5 | 1 | 0 | 0

2. Secondary Outcome: Overall Response Rate
Description: Overall response rate by International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria following 6 months of biweekly dosing of cirmtuzumab
Time Frame: From start of investigational treatment to discontinuation from trial participation, on average 159 days
Measure: Number; unit: percentage of participants
Arm/Group | Cirmtuzumab
Number analyzed (Participants) | 3
percentage of participants | 0

3. Secondary Outcome: Progression Free Survival (PFS)
Description: The duration of time from the start of study treatment until objective tumor progression or death determined by International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria
Time Frame: From start of investigational treatment to tumor progression or death, on average 16.66 months
Population: Only one subject progressed after being on study at 16.66 months. The other two subjects did not progress but went off study at months 3.84 and 1.26, respectively; thus, their PFS status was censored at off study date.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Cirmtuzumab
Number analyzed (Participants) | 1
months | 16.66 (0)

4. Secondary Outcome: Stable Disease Rate (SD)
Description: The Stable Disease Rate based on number of subjects who have absence of disease progression as determined by International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria.
Time Frame: From start of investigational treatment to discontinuation from trial participation, on average 159 days
Measure: Number; unit: percentage of participants
Arm/Group | Cirmtuzumab
Number analyzed (Participants) | 3
percentage of participants | 100

5. Secondary Outcome: Partial Response Rate (PR)
Description: The percentage of subjects who achieve partial clinical response determined by International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria.
Time Frame: From start of investigational treatment to discontinuation from trial participation, on average 159 days
Population: All 3 patients has stable disease while on treatment. Partial response rate is therefore 0%.
Measure: Number; unit: percentage of participants
Arm/Group | Cirmtuzumab
Number analyzed (Participants) | 3
percentage of participants | 0

6. Secondary Outcome: Undetectable Minimal Residual Disease (uMRD) Rate
Description: The Undetectable Minimal Residual Disease rate based on the number of subjects achieving undetectable minimal residual disease as determined by International Workshop on Chronic Lymphocytic Leukemia (iWCLL) criteria.
Time Frame: From start of investigational treatment to discontinuation from trial participation, on average 159 days
Measure: Number; unit: percentage of participants
Arm/Group | Cirmtuzumab
Number analyzed (Participants) | 3
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during treatment with cirmtuzumab and during the post-treatment follow-up period until the last subject's discontinuation from trial participation, on average 159 days.
Arm/Group | Cirmtuzumab
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cirmtuzumab (N=3)
Eye disorders, other (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders, other (Gastrointestinal disorders) | 1 (1)
Dizziness (General disorders) | 1 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Anemia (Investigations) | 3 (6)
Thrombocytopenia (Investigations) | 3 (7)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders, other (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/76/NCT02860676/Prot_SAP_000.pdf